CLINICAL TRIAL: NCT03038958
Title: Comparison of Hyperbaric Prilocaine With Chloroprocaine for Intrathecal Anaesthesia in Day Case Knee Arthroscopy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Saint Pierre (Other)
Collaborators: Hôpital de Braine-l'Alleud (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AK160324627AD
Record Dates: First submitted 2017-01-26; First posted 2017-02-01 (Estimated); Last update posted 2019-11-18 (Actual); Status verified 2019-11

CONDITIONS: Knee Arthroscopy; Spinal Anesthesia
Keywords: Local Anaesthetic; spinal anesthesia; Knee arthroscopy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Isobaric 2-chloroprocaine (Active Comparator): The 50 mg dose of isobaric 2-chloroprocaine will be administered to patients undergoing ambulatory knee arthroscopy
  Interventions: Drug: Isobaric 2-chloroprocaine
- Hyperbaric prilocaine 2% (Active Comparator): The dose of 50 mg of Hyperbaric prilocaine 2% will be administered to patients undergoing ambulatory knee arthroscopy
  Interventions: Drug: Hyperbaric prilocaine

INTERVENTIONS:
Drug: Isobaric 2-chloroprocaine — intrathecal injection of 50 mg isobaric 2-Chloroprocaine
  Other Names: Ampres
  Arms: Isobaric 2-chloroprocaine
Drug: Hyperbaric prilocaine — intrathecal injection of 50 mg hyperbaric prilocaine 2%
  Other Names: Tachipri
  Arms: Hyperbaric prilocaine 2%

SUMMARY:
This study compares intrathecal 1% plain chloroprocaine with intrathecal 2% hyperbaric prilocaine for patients undergoing ambulatory knee arthroscopy in terms of efficacy and side effects

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiology physical status (ASA) ≤ III
* Age 18-80 year
* Height between 160 and 185 cm
* Signed informed consent obtained prior to any study specific assessments and procedures

Exclusion Criteria:

* Cardiac pathology (such as Heart failure, Aortic stenosis)
* Coagulation disorders (INR>1.3, platelet < 80 000/mm3)
* Known allergy to local anaesthetics
* Disagreement of the patient

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2016-04; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Duration of sensory block | Until complete release of sensory block
  Total duration of sensory block is the interval time between the end of intrathecal injection and the complete recovery of sensory block

SECONDARY OUTCOMES:
Onset time of sensory block | up to 30 minutes
  The levels of sensory block will be determined at 5, 10, 20 and 30 minutes after intrathecal injection. The levels of sensory block will be assessed as loss of sensation to pin-prick and cold.
Onset time of motor block | up to 30 minutes
  The levels of motor block will be determined at 5, 10, 20 and 30 minutes after intrathecal injection. The levels of motor block will be assessed by using the Bromage Scale (0=no motor block; 1=hip blocked; 2=hip and knee blocked; 3=hip, knee, and ankle blocked).
Duration of motor block | Until complete regression of motor block
  Total duration of motor block is the interval time between the end of intrathecal injection and the complete recovery of motor block
Pain assessed by Visual Analog Scale | up to 24 hours
  Pain levels will be determined at the inflation of tourniquet, at the incision and every 10 minutes in the PACU (Post Anesthesia Care Unit). Visual Analog pain score (scale = 0 no pain; 10 = worst pain imaginable).
Side-effects (hypotension, bradycardia, urinary retention) | up to 24 hours
  Assessed during and after intervention

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel Guntz, MD, Study Director — Université Libre de Bruxelles (ULB), Braine-l'Alleud Hospital; Panayota Kapessidou, MD,PhD, Principal Investigator — University Hospital Saint-Pierre (CHU Saint-Pierre), Université Libre de Bruxelles (ULB)
Locations (2):
- Belgium (2):
  - Braine-l'Alleud Hospital, Braine-l'Alleud
  - CHU Saint-Pierre, Brussels Capital Region

IPD SHARING:
Plan to Share IPD: No